CLINICAL TRIAL: NCT02444949
Title: A Trial of Endostar in Combination With Chemotherapy of DF and Sequential Intensity Modulated Radiation Therapy for Patients With Advanced Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Three Gorges University, Yichang, China (Other)
Responsible Party: Principal Investigator, Xin-Hua Xu, The section chief of Oncology Department, The First College of Clinical Medical Science, China Three Gorges University, China Three Gorges University, Yichang, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTGU001
Record Dates: First submitted 2015-04-07; First posted 2015-05-15 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — endostar protein; Cisplatin

ARMS (2):
- endostar+DF+IMRT (Experimental): patient first receive one periodicity chemotherapy(DDP (25mg/m2/d; ivgtt; d1～3)+5-FU (600mg/m2/d; ivgtt; d1～5)+endostar (150mg/5d; civ; d1～5)), then given IMRT (5 times per week, 6 weeks). After rest 4 weeks, continue to give the chemotherapy (21 days for a periodicity, 3 periodicities).
  Interventions: Drug: endostar; Radiation: intensity modulated radiation; Drug: cisplatin
- DF+IMRT (Other): patient first receive one periodicity chemotherapy(DDP (25mg/m2/d; ivgtt; d1～3)+5-FU (600mg/m2/d; ivgtt; d1～5)), then given IMRT (5 times per week, 6 weeks). After rest 4 weeks, continue to give the chemotherapy (21 days for a periodicity, 3 periodicities).
  Interventions: Radiation: intensity modulated radiation; Drug: cisplatin

INTERVENTIONS:
Drug: endostar
  Other Names: Human recombinant vascular endothelial inhibitor
  Arms: endostar+DF+IMRT
Radiation: intensity modulated radiation
Drug: cisplatin
  Other Names: DDP

SUMMARY:
Among all the head and neck tumors, nasopharyngeal carcinoma (NPC) has a high tendency of recurrence and metastasis. For the advanced NPC patients, chemoradiotherapy is the main way of treatment. Currently, chemotherapy with cisplatin (DDP) combines with 5-fluorouracil (5-FU) is the classic front line therapy for NPC. However, the abnormal richness of angiogenesis of tumor and blood supply in tissue caused by radiation therapy often decrease the effects of radiochemotherapy. Human recombinant vascular endothelial inhibitor (endostar) can improve the sensitivity to chemoradiation via selectively inhibiting the migration of endothelial cells and the formation of tumor vessels. Moreover, it would induce vascular remodeling and normalization of the tumor vasculature, which will effectively aid the delivery of oxygen and anticancer drugs. In sum, antiangiogenesis in combination with chemoradiotherapy will be a promising way of treatment for NPC. In this study, the first-treated patients with NPC (stage Ⅲ or Ⅳa) confirmed by pathology, and patients with recurrent and metastatic NPC will be randomly assigned to two groups (1:1): a trial group (DDP, 5-FU, endostar and sequential intensity modulated radiation therapy (IMRT)), and a control group (DDP，5-FU and sequential IMRT). Evaluations will be developed including progression-free survival (PFS), Overall response rate（ORR）, overall survival (OS), adverse effects rate and quality of life. This research will provide more evidences of evidence-based medicine for the safety and tolerability of endostar and the clinical application of endostar in NPC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 ears ;
* Eastern Cooperative Oncology Group performance status of 0-1;
* diagnosed with first-treated NPC (Ⅲ/Ⅳa stage) confirmed by pathology;
* ecurrent and metastatic NPC with indication of chemoradiotherapy;
* one measurable lesion at least (according to the RECIST guidelines, the lesion iameter≥20 mm with MRI);
* life expectancy of ≥ 12 weeks;
* adequate hematologic, renal, cardiac and liver function;
* hemameba≥4.0×109/L;
* neutrophil≥2.0×109/L;
* platelet≥100×109/L;
* hemoglobin≥95g/L;
* Serum bilirubin, ALT and AST ≤1.5 times of maximum criteria;
* sufficiently understand this study situation and signed the informed consent.

Exclusion Criteria:

* allergy or intolerance to study drugs;
* receiving other anti-cancer therapy;
* uncontrolled central nervous system lesions;
* dysfunction of important organs；
* history of cardiovascular disease(including congestive heart-failure, uncontrolled arrhythmia, angina pectoris which require long-term drug treatment, lular heart disease, myocardial infarction and resistant hypertension);
* pregnancy or lactation in women;
* protracted Infective wound;
* history of mental illness which is not easy controlled.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | Patients will be followed from the day in which patients are enrolled the clinical trial and end up one year later, during the one year the patients will be observed whether they have disease progress or die from any cause.
Overall response rate | After the second periodicity chemotherapy, an expected average of 12 weeks, the rate of patients with complete response and partial response accounted for the total number of assessable cases .

SECONDARY OUTCOMES:
Adverse effects as assessed by adverse events | It is the time from the start of treatment to 20 weeks
Overall survival | Patients will be followed from the day in which patients are enrolled the clinical trial and end up two years later, during the two years the patients will be observed whether they die from any cause.
Quality of Life measured by the ECDG score | Firstly, Patients will be assessed before the start of periodicity treatment, then they will be assessed 20 weeks and 24 weeks after the treatment.